CLINICAL TRIAL: NCT02629796
Title: Biomarker to Predict the Response to Intravenous Immunoglobulin in Chronic Inflammatory Demyelinating Polyradiculoneuropathy Patients: a Transcriptomic Study
Brief Title: Biomark Study: Predict Intravenous Immunoglobulin Responders in Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Acronym: BIOMARK
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AGN_2013-9
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: CIDP
Keywords: Biomarker; CIDP; IVIG; treatment response
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- CIDP treated (IVIG): patients with a diagnosis of chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) according to European criteria, treated with IVIG (intravenous immunoglobulin as a first line of treatment) as a usual treatment
  Interventions: Other: CIDP treated (IVIG)
- control: healthy subjects

INTERVENTIONS:
Other: CIDP treated (IVIG) — usual treatment with intravenous immunoglobulin
  Groups: CIDP treated (IVIG)

SUMMARY:
This study aims analyze the transcriptome to identify predictive biomarkers of IVIG in CIDP patients. 25 patients with a diagnosis of CIDP according to European criteria, naïve of treatment, will be included and followed for 1 year. Clinical assessment (RT-MRC ; Martin vigorimeter, RT-mISS,R-ODS,TW25, 9hole-peg test) will be performed at baseline and at 3, 6 and 12 months after the first IVIG course. Responder/No responder status will be defined at 3 month and confirmed at 12 months. Blood samples will be collected before the IVIG course at baseline, and at 2months and 6 months. At the end of the first IVIG course a blood sample will be collected to assess early changes of transcriptome. The CIDP diagnosis and responder/no responder status will be confirmed by an independent committee. The transcriptome of the patients will be individually analyzed and compared regarding Responder/Non responder status to a control groups of 20 healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* chronic inflammatory demyelinating polyradiculoneuropathy (according to european criterions)
* first line of treatment
* treatment with intravenous immunoglobulin required
* healthy subjects matched for age and gender

Exclusion Criteria:

For CIDP patients

* uncontrolled diabetes, monoclonal spike with anti-ganglioside activity, anti myelin-associated glycoprotein antibodies, HIV infection, HBV infection, HCV infection, connective tissue disease, hemopathy, evolutive disease)

For healthy subjects:

any chronic or autoimmune disease

For all subjets viral or bacterial infection in the last 30 days chemotherapy in the last 5 years immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with chronic inflammatory demyelinating polyradiculoneuropathy. Transcriptome, metabolome and proteome analysis compared with those of healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2014-04-16 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
blood-levels of biomarkers of Intravenous immunoglobulin response | 8 weeks

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU Bordeaux, service de Neurologie, Bordeaux, Aquitaine
  - CHU Nantes, Laboratoire d'explorations fonctionnelles, Nantes, Loire Atlantique
  - CHU de Brest, Brest
  - CHU de CAEN, Caen
  - Service de Neurologie Hopital du Kremlin Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - Service de Neurologie, CHU Limoges,, Limoges
  - Hôpital Neurologique HCL, Lyon-Bron, Lyon
  - CHU de NIMES, Nîmes
  - Service de Physiologie Clinique - Explorations Fonctionnelles, Hôpital Lariboisière, Paris
  - Service de Neurologie, Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Centre Hospitalier Intercommunal de Poissy/Saint-Germain-en-Laye, Poissy
  - CHU de Poitiers, Poitiers
  - CHU de ROUEN, Rouen
  - Centre Hospitalier de Saint-Denis, Saint-Denis
  - Service de Neurologie CHU St Etienne, Saint-Etienne
  - Service de Neurologie, CHU de Strasbourg, Strasbourg
  - CHU Henri Mondor, Créteil, Île-de-France Region